CLINICAL TRIAL: NCT04618822
Title: Motor-enriched Learning for Improving Pre-reading and Word Recognition Skills in Preschool Children Aged 5-6 Years
Brief Title: Play-based Motor-Cognitive Training for Improved Reading
Acronym: PLAYMORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jacob Wienecke, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8018-00132B
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Reading
Keywords: motor-enriched learning; embodied learning; physically active lessons; pre-reading skills; word recognition; preschool children

STUDY DESIGN:
Intervention Model Description: A three-armed randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teaching involving whole-body movements (Experimental)
  Interventions: Behavioral: Teaching involving whole-body movements
- Teaching involving hand movements (Experimental): i.e. arms and hands
  Interventions: Behavioral: Teaching involving hand movements
- teaching involving minimal motor movements (Active Comparator): i.e. seated on a chair using paper and pencil
  Interventions: Behavioral: Teaching involving minimal motor movements (control)

INTERVENTIONS:
Behavioral: Teaching involving whole-body movements — The intervention consist of three 30 minutes sessions per week for eight weeks. Activities are conducted in small groups of six children and focus on the acquisition of letterforms, letter-sound correspondences and reading and spelling of short words. Activities involve whole-body movements and have been developed with the embodied learning theory in mind, linking movement closely to the learning content.
  Arms: Teaching involving whole-body movements
Behavioral: Teaching involving hand movements — The intervention consist of three 30 minutes sessions per week for eight weeks. Activities are conducted in small groups of six children and focus on the acquisition of letterforms, letter-sound correspondences and reading and spelling of short words. Activities involve movements using hands and arms and have been developed with the embodied learning theory in mind, linking movement closely to the learning content.
  Arms: Teaching involving hand movements
Behavioral: Teaching involving minimal motor movements (control) — The control condition consist of three 30 minutes sessions per week for eight weeks. Activities are conducted in groups of app. twelve children and focus on the acquisition of letterforms, letter-sound correspondences and reading and spelling of short words. Activities are completed seated on a chair using paper and pencil.
  Arms: teaching involving minimal motor movements

SUMMARY:
The PLAYMORE study aims to investigate the effects of two interventions focusing on a close and meaningful coupling between bodily movement and academic content on early pre-reading and word recognition skills in children. Further, the study aims to compare two interventions involving either hand movements (i.e. using arms and hands) or whole-body movements (i.e. using the whole body). Potential mediating factors underlying the potential effect of bodily movement on early pre-reading and word recognition skills will be explored. The PLAYMORE study will be conducted as a three-armed randomized controlled trial including children aged five to six years recruited from four schools in the Copenhagen area, Denmark. Stratified by class, children will be randomly allocated to one of three 8-week intervention/control periods: 1) teaching involving whole-body movements, 2) teaching involving hand movements (i.e. arms and hands) or 3) teaching involving minimal motor movements (i.e. seated on a chair using paper and pencil). Outcome measurements, including pre-reading and word recognition skills, will be collected before and after the intervention period to assess the intervention effects. This study protocol follows the SPIRIT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Children five to six years old who have just started school

Exclusion Criteria:

* Children who do not speak any Danish
* Children with cognitive or physical disabilities hindering participation in the project activities

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in word reading speed and accuracy (reading of 18 trained words) at 8 weeks, computer-based test | Baseline and 8-weeks
  This word reading test consist of 18 presentations of targets words; one target word per presentation. Below the target word are placed four pictures of which one illustrates the target word. For the children to give a correct answer, they will have to touch the picture matching the target word on the touch screen. They are asked to touch the correct picture as fast as possible. The three remaining pictures represents words (distractors) that have either the initial (two pictures) or the final (one picture) sound in common with the target word. The presentations of target words and the order of the four pictures are randomized between subjects and time points. During the test, children are allowed to ask questions concerning the pictures (e.g. what is shown on this picture?) but not regarding the target word (e.g. what is the sound of this letter?). The results from the test constitute mean response time for correct answers and number of correct answers.
Change from baseline in trained letter-sound correspondences accuracy (15 trials) at 8 weeks, paper and pencil test | Baseline and 8-weeks
  The test consists of 15 trials. In each trial, a sound corresponding to a standard or a conditional pronunciation of a letter is said out loud by the assessor. Children are instructed to identify the correct letter matching the sound from a row of four letters. Before the test trials, children will be provided with one practice trial. The 15 sounds represent both standard and conditional pronunciations of the letters a, e, o, r, u and v. Results are numbers of correct letter-sound correspondences.

SECONDARY OUTCOMES:
Change from baseline in word reading accuracy (reading of 12 untrained words) at 8 weeks, computer-based test | Baseline and 8-weeks
  This test consists of 12 presentations of untrained words; one word per presentation. The 12 words consist of four 2-letter words, four 3-letter words and four 4-letter words.
Change from baseline in letter naming fluency accuracy at 8 weeks | Baseline and 8-weeks
  This Danish version of the Letter Naming test is based on the same principles as DIBELS Letter Naming Fluency (Good & Kaminski, 2002). The test consists of a piece of paper (A4) with 12 rows of 10 letters (mixed upper- and lower case).
Change from baseline in letter-sound correspondence accuracy, Bogstaveprøve 2 ['Letter test 2'] at 8 weeks | Baseline and 8-weeks
  This test has been widely used in the Danish school system. The test consists of two subtests assessing simple letter-sound knowledge and vowel identification, respectively. For the purpose of the present study, only the first subtest will be administered to assess standard letter-sound knowledge.
Change from baseline in word reading accuracy and speed, Ordlæseprøve 1 ['Word reading test 1'] at 8 weeks | Baseline and 8-weeks
  This test is widely used in the Danish school system. The test consists of 78 items (preceded by two practice items) and evaluates word reading accuracy as well as efficiency.
Change from baseline in word reading speed and accuracy (reading of 18 trained words) at 18 weeks, computer-based test | Baseline and 18-weeks
  This word reading test consist of 18 presentations of targets words; one target word per presentation. Below the target word are placed four pictures of which one illustrates the target word. For the children to give a correct answer, they will have to touch the picture matching the target word on the touch screen. They are asked to touch the correct picture as fast as possible. The three remaining pictures represents words (distractors) that have either the initial (two pictures) or the final (one picture) sound in common with the target word. The presentations of target words and the order of the four pictures are randomized between subjects and time points. During the test, children are allowed to ask questions concerning the pictures (e.g. what is shown on this picture?) but not regarding the target word (e.g. what is the sound of this letter?). The results from the test constitute mean response time for correct answers and number of correct answers.
Change from baseline in trained letter-sound correspondences accuracy (15 trials) at 18 weeks, paper and pencil test | Baseline and 18-weeks
  The test consists of 15 trials. In each trial, a sound corresponding to a standard or a conditional pronunciation of a letter is said out loud by the assessor. Children are instructed to identify the correct letter matching the sound from a row of four letters. Before the test trials, children will be provided with one practice trial. The 15 sounds represent both standard and conditional pronunciations of the letters a, e, o, r, u and v. Results are numbers of correct letter-sound correspondences.
Change in word reading speed and accuracy (reading of 18 trained words) between 8 weeks and 18 weeks, computer-based test | 8-weeks and 18-weeks
  This word reading test consist of 18 presentations of targets words; one target word per presentation. Below the target word are placed four pictures of which one illustrates the target word. For the children to give a correct answer, they will have to touch the picture matching the target word on the touch screen. They are asked to touch the correct picture as fast as possible. The three remaining pictures represents words (distractors) that have either the initial (two pictures) or the final (one picture) sound in common with the target word. The presentations of target words and the order of the four pictures are randomized between subjects and time points. During the test, children are allowed to ask questions concerning the pictures (e.g. what is shown on this picture?) but not regarding the target word (e.g. what is the sound of this letter?). The results from the test constitute mean response time for correct answers and number of correct answers.
Change in trained letter-sound correspondences accuracy (15 trials) between 8 weeks and 18 weeks, paper and pencil test | 8-weeks and 18-weeks
  The test consists of 15 trials. In each trial, a sound corresponding to a standard or a conditional pronunciation of a letter is said out loud by the assessor. Children are instructed to identify the correct letter matching the sound from a row of four letters. Before the test trials, children will be provided with one practice trial. The 15 sounds represent both standard and conditional pronunciations of the letters a, e, o, r, u and v. Results are numbers of correct letter-sound correspondences.
Change in word reading accuracy (reading of 12 untrained words) between 8 weeks and 18 weeks, computer-based test | 8-weeks and 18-weeks
  This test consists of 12 presentations of untrained words; one word per presentation. The 12 words consist of four 2-letter words, four 3-letter words and four 4-letter words.
Change in letter naming fluency accuracy between 8 weeks and 18 weeks | 8-weeks and 18-weeks
  This Danish version of the Letter Naming test is based on the same principles as DIBELS Letter Naming Fluency (Good & Kaminski, 2002). The test consists of a piece of paper (A4) with 12 rows of 10 letters (mixed upper- and lower case).
Change in letter-sound correspondence accuracy, Bogstaveprøve 2 ['Letter test 2'] between 8 weeks and 18 weeks | 8-weeks and 18-weeks
  This test has been widely used in the Danish school system. The test consists of two subtests assessing simple letter-sound knowledge and vowel identification, respectively. For the purpose of the present study, only the first subtest will be administered to assess standard letter-sound knowledge.
Change in word reading accuracy and speed, Ordlæseprøve 1 ['Word reading test 1'] between 8 weeks and 18 weeks | 8-weeks and 18-weeks
  This test is widely used in the Danish school system. The test consists of 78 items (preceded by two practice items) and evaluates word reading accuracy as well as efficiency.

OTHER OUTCOMES:
Change in 1-back task accuracy and reaction time | Baseline, 8-weeks and 18-weeks
  This 1-back task is constructed of representations of symbols (car, cloud, globe, note, headphones, airplane, plate, key, eye and bicycle); one symbol is presented at the time.
Change in digit span forwards and backwards accuracy (number of correctly remembered sequences and the number of digits in the longest correctly remembered sequence) | Baseline, 8-weeks and 18-weeks
  The digit span task is a subtest of the Wechsler Intelligence Scale for Children - fourth edition (WISC-IV) (Wechsler, 2003) and is used to assess auditory working memory, attention, and concentration. The test consists of two subtests; digit span forward and digit span backwards.
Intrinsic motivation questionnaire | Four times during study completion, immediately after one session in week two, four, six and eight
  Modified version of Intrinsic Motivation Inventory (IMI) (McAuley, Duncan, & Tammen, 1989). The original items of the IMI are translated into Danish using a translation-backtranslation process (Streiner & Norman, 2008). The inventory is reduced to six questions related to intrinsic motivation (question 1-3) and feeling of competences (question 4-6).
Change in Flamingo balance test, balance on one leg (sum of attempts with both legs; lower scores indicate better performance) | Baseline, 8-weeks and 18-weeks
  The flamingo balance test is a standardized test that assesses the ability to balance successfully on one leg (Adam, C., Klissouras, V., Ravazzolo, M., Renson, R., & Tuxworth, 1988).
Change in 9-hole pegboard (speed) | Baseline, 8-weeks and 18-weeks
  The 9-hole pegboard test is a standardized test which has previously been used in children to evaluate fine motor skills (Longcamp et al., 2005; Smith, Hong, & Presson, 2000).
Flamingo balance test, balance on one leg (sum of attempts with both legs; lower scores indicate better performance) | Baseline
  The flamingo balance test is a standardized test that assesses the ability to balance successfully on one leg (Adam, C., Klissouras, V., Ravazzolo, M., Renson, R., & Tuxworth, 1988).
9-hole pegboard (speed) | Baseline
  The 9-hole pegboard test is a standardized test which has previously been used in children to evaluate fine motor skills (Longcamp et al., 2005; Smith, Hong, & Presson, 2000).
Letter-sound correspondence accuracy, Bogstaveprøve 2 ['Letter test 2'] | Baseline
  This test has been widely used in the Danish school system. The test consists of two subtests assessing simple letter-sound knowledge and vowel identification, respectively. For the purpose of the present study, only the first subtest will be administered to assess standard letter-sound knowledge.
Word reading accuracy and speed, Ordlæseprøve 1 ['Word reading test 1'] | Baseline
  This test is widely used in the Danish school system. The test consists of 78 items (preceded by two practice items) and evaluates word reading accuracy as well as efficiency.
Letter naming fluency accuracy | Baseline
  This Danish version of the Letter Naming test is based on the same principles as DIBELS Letter Naming Fluency (Good & Kaminski, 2002). The test consists of a piece of paper (A4) with 12 rows of 10 letters (mixed upper- and lower case).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gejl AK, Malling ASB, Damsgaard L, Veber-Nielsen AM, Wienecke J. Motor-enriched learning for improving pre-reading and word recognition skills in preschool children aged 5-6 years - study protocol for the PLAYMORE randomized controlled trial. BMC Pediatr. 2021 Jan 4;21(1):2. doi: 10.1186/s12887-020-02430-0. PMID 33397297